CLINICAL TRIAL: NCT00725517
Title: Efficacy and Safety of a 7.5% Icodextrin Peritoneal Dialysis Solution in Once-Daily Long Dwell Exchange in Continuous Ambulatory Peritoneal Dialysis Patients, Compare to 2.5% Dianeal Peritoneal Dialysis Solution.
Brief Title: Efficacy and Safety of a 7.5% Icodextrin Peritoneal Dialysis Solution in Once-Daily Long Dwell Exchange
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Jiaqi Qian, renji hospital, shanghai jiaotong university school of medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN-R-001
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Kidney Disease; Peritoneal Dialysis
Keywords: Icodextrin; ultrafiltration; creatinine clearance; urea nitrogen clearance
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Icodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Icodextrin group
  Interventions: Drug: Icodextrin
- 2 (No Intervention): Glucose group

INTERVENTIONS:
Drug: Icodextrin — Icodextrin was used instead of Dianeal for long dwell time every day for 5 weeks.
  Other Names: Extraneal dialysate
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a 7.5% Icodextrin peritoneal dialysis solution for once-daily long dwell exchange in patients undergoing Continuous Ambulatory Peritoneal Dialysis (CAPD) in Chinese uremic patients.Patients were divided into Dianeal group or Extraneal group for long dwell time. Net ultrafiltration, small solute clearance and relationship between different transport group were used to evaluate efficacy of Icodextrin. Physical examination, vital signs and laboratory tests were used to evaluate safety of Icodextrin.

DETAILED DESCRIPTION:
A prospective, multicenter, randomized, double blind, parallel controlled study has been conducted for 5 weeks in 201 CAPD patients. These patients were randomized from 7 centers with 98 allocated to the Icodextrin group and 103 to the Dextrose group. Before study, conventional glucose-based solution was the only dialysate which can available in China. Extraneal® is one of peritoneal dialysate produced by Baxter which contains 7.5% Icodextrin. Patients involved the study were allocated to Dianeal group and Extraneal group in randomize. In Dianeal group, prescription was unchanged, while in Extraneal group, Extraneal dialysate was used instead of 2.5% Dianeal. Assessments at baseline, week 2, and week 4 included drain volume and levels of glucose, creatinine, and urea in the dialysate drained from the long dwell; physical examination; vital signs; drained body weight; laboratory analyses. Daily net peritoneal ultrafiltration, daily peritoneal creatine clearance and daily peritoneal urea nitrogen clearance were recorded prior to and 2 week, 4 week after commencing Extraneal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing continuous ambulatory peritoneal dialysis (CAPD) for more than 90 days were included in the study.
2. Over the age of 18
3. Received a minimum of 6-8 liters of dialysis fluid per day and nighttime must lasted for 8-16 hours with 2.5% Dianeal® PD-2 or PD-4 dialysate, dwell volume was 2.0 liters before 30 days of screen visit
4. No acute/chronic exit infection or tunnel infection accompany with peritonitis infection before 30 days of screen visit

Exclusion Criteria:

1. Be sensitive to Icodextrin
2. Suffer from other serious disease
3. Attended other invention research which was approved by Ethics Committee
4. Used other drugs in trial 30 days before screen visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
long dwell net peritoneal ultrafiltration | 5 weeks

SECONDARY OUTCOMES:
long dwell peritoneal creatine clearance and long dwell peritoneal urea nitrogen clearance, physical examination; vital signs; drained body weight; laboratory analyses | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqi Qian, MD, Principal Investigator — RenJi Hospital